CLINICAL TRIAL: NCT04417127
Title: Harambee: Integrated Community-based HIV/NCD Care & Microfinance Groups in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Johns Hopkins University (Other); Moi University (Other); Purdue University (Other); University of Toronto (Other); NYU Langone Health (Other); Academic Model Providing Access to Healthcare (AMPATH) (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Omar Galarraga, PhD, ASSOCIATE PROFESSOR, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH118075 (NIH); R01MH118075 (NIH)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: HIV/AIDS; Noncommunicable Diseases; Hypertension; Diabetes
Keywords: HIV, Noncommunicable Diseases, microfinance, differentiated care, mobile care, telemedicine, task-shifting
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Noncommunicable Diseases; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Aim 1: Cluster randomized trial where a minimum of 40 existing microfinance groups with n=900 members are randomized 1:1 to receive either integrated community-based care (ICB) or usual care. Delivered quarterly during community-based microfinance meetings, the intervention includes: clinical consultations, diabetes and/or hypertension management, distribution of antiretroviral therapy and NCD medications, health education, and facility referrals. Members of microfinance groups randomized to usual care will continue to receive care at a health facility. Aim 1 will also enroll an additional n=300 frequency-matched, prospectively-followed usual care patients without microfinance. Aim 2: Mediation analyses with n=40 trial participants and n=10 intervention staff. Aim 3: Cost-effectiveness analyses with n=5 budget staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microfinance with Integrated Community-based Care (Experimental): A minimum of 20 microfinance groups with approximately n=450 participants will be randomized to receive the ICB intervention.
  Interventions: Other: Integrated Community-Based (ICB) Care; Other: Group-level Microfinance
- Microfinance with Usual (Facility-Based) Care (Active Comparator): A minimum of 20 microfinance groups with approximately n=450 participants will be randomized to continue to receive standard of care from an AMPATH-supported rural health facility.
  Interventions: Other: Group-level Microfinance
- Usual (Facility-Based) Care without Microfinance (No Intervention): A total of n=300 participants who receive care at an AMPATH health facility and who are not involved in microfinance will serve as frequency-matched contemporaneous controls. These participants will be actively followed over the 18-months of the trial.

INTERVENTIONS:
Other: Integrated Community-Based (ICB) Care — During quarterly intervention visits, a clinical officer (CO) travels to the location of the microfinance group meeting. The CO meets privately with each patient one-on-one, provides brief medical consultations, and distributes ART and other medications for diabetes and hypertension as needed. ART medicines are provided at no cost to patients from AMPATH HIV pharmacies; medications for diabetes and hypertension are dispensed to patients from AMPATH Revolving Fund Pharmacies at a standardized price. The CO conducts point-of-care laboratory testing if medically indicated. Every 6 months, the CO conducts a more intensive HIV clinical evaluation. The cost of point-of-care tests administered at study baseline and study end line are covered by the study. Additional tests during the trial are paid for by the patient. COs make referrals to facilities for emergency or acute care needs. Each visit includes a health education discussion conducted in a group.
  Arms: Microfinance with Integrated Community-based Care
Other: Group-level Microfinance — Group microfinance uses a client-driven model that involves community savings groups where members mobilize and manage their own savings, provide interest-bearing loans to group members, offer a limited form of financial insurance, and contribute to a social fund that is used for income-generating activities and in cases of emergency or welfare issues of group members.
  For this study, group microfinance will refer to existing, active AMPATH Group Integrated Savings for Empowerment (GISE) microfinance groups with a majority of group members who are AMPATH HIV patients and have disclosed their HIV status. Groups will be considered active if the group was formed at least 6 months prior to study baseline, is consistently meeting as scheduled, and is actively engaging in saving and loaning.
  Arms: Microfinance with Integrated Community-based Care; Microfinance with Usual (Facility-Based) Care

SUMMARY:
The objective of this project is to demonstrate the effectiveness and longer-term sustainability of a differentiated care delivery model for improving HIV treatment outcomes. The central hypothesis is that the integration of community-based HIV and NCD care with group microfinance will improve retention in care and rates of viral suppression (VS) among people living with HIV (PLHIV) in Kenya via two mechanisms: improved household economic status and easier access to care.

The specific aims are as follows:

1. To evaluate the extent to which integrated community-based HIV care with group microfinance affects retention in care and viral suppression among n=900 PLHIV in rural western Kenya using a cluster randomized intervention design of at least n=40 existing (fully HIV+) microfinance groups to receive either: (A) integrated community-based HIV and NCD care or (B) usual facility-based care. Data from the two trial arms will be augmented with a matched contemporaneous control group of n=300 patients receiving usual facility-based care and not involved in microfinance (group C), comparing outcomes in groups A, B and C. The hypothesize is that A > B > C in terms of viral suppression and retention in care.
2. To identify specific mechanisms through which microfinance and integrated community-based care impact viral suppression. Using a mixed methods approach, the study will characterize the mechanisms of effect on patient outcomes. Investigators will conduct quantitative mediation analysis to examine two main mediating pathways (household economic conditions and easier access to care), as well as exploratory mechanisms (food security, social support, HIV- related stigma). Investigators will also use qualitative methods and multi-stakeholder panels to contextualize implementation of the intervention.
3. To assess the cost-effectiveness of microfinance and integrated community-based care delivery to maximize future policy and practice relevance of this promising intervention strategy. The working hypothesis is that the differentiated model will be cost-effective in terms of cost per HIV suppressed person-time, cost per patient retained in care, and cost per disability-adjusted life year saved.

The main expected outcomes will be rigorous evidence of effectiveness, mechanisms and cost-effectiveness of a differentiated model for achieving the last key step in the HIV care continuum. These results are expected to have an important positive impact in terms of improved, high-quality services that address known individual and structural barriers to care and promote long-term sustainability of care for PLHIV in rural settings with high HIV prevalence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at study baseline
* HIV-positive
* Have received any care through AMPATH since 2010
* Initiated ART at least 6 months prior to study baseline
* Have participated in at least one microfinance group meeting in the prior 12 months at study baseline (for Study Arms A & B)
* Willing and able to provide informed consent.

Exclusion Criteria:

* Currently participating in the BIGPIC study
* Unable to provide informed consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University/ Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No
Materials generated under this project will be disseminated according to University and NIH policies regarding data sharing. Aggregate-level data collected in this collaboration will ultimately be available for public use. Opportunities for secondary analyses will be available following completion of the three-year project and publication of the main study findings. These findings will be available to the public through scientific meetings and peer-reviewed journals, as well as through a structured policy dissemination process.

REFERENCES:
- [Background] Kafu C, Wachira J, Omodi V, Said J, Pastakia SD, Tran DN, Onyango JA, Aburi D, Wilson-Barthes M, Galarraga O, Genberg BL. Integrating community-based HIV and non-communicable disease care with microfinance groups: a feasibility study in Western Kenya. Pilot Feasibility Stud. 2022 Dec 28;8(1):266. doi: 10.1186/s40814-022-01218-6. PMID 36578093
- [Background] Genberg BL, Wilson-Barthes MG, Omodi V, Hogan JW, Steingrimsson J, Wachira J, Pastakia S, Tran DN, Kiragu ZW, Ruhl LJ, Rosenberg M, Kimaiyo S, Galarraga O. Microfinance, retention in care, and mortality among patients enrolled in HIV care in East Africa. AIDS. 2021 Oct 1;35(12):1997-2005. doi: 10.1097/QAD.0000000000002987. PMID 34115646
- [Background] Genberg BL, Wachira J, Steingrimsson JA, Pastakia S, Tran DNT, Said JA, Braitstein P, Hogan JW, Vedanthan R, Goodrich S, Kafu C, Wilson-Barthes M, Galarraga O. Integrated community-based HIV and non-communicable disease care within microfinance groups in Kenya: study protocol for the Harambee cluster randomised trial. BMJ Open. 2021 May 18;11(5):e042662. doi: 10.1136/bmjopen-2020-042662. PMID 34006540
- [Background] Tran DN, Ching J, Kafu C, Wachira J, Koros H, Venkataramani M, Said J, Pastakia SD, Galarraga O, Genberg BL. Interruptions to HIV Care Delivery During Pandemics and Natural Disasters: A Qualitative Study of Challenges and Opportunities From Frontline Healthcare Providers in Western Kenya. J Int Assoc Provid AIDS Care. 2023 Jan-Dec;22:23259582231152041. doi: 10.1177/23259582231152041. PMID 36718505
- [Background] Wilson-Barthes M, Steingrimsson J, Lee Y, Tran DN, Wachira J, Kafu C, Pastakia SD, Vedanthan R, Said JA, Genberg BL, Galarraga O. Economic outcomes among microfinance group members receiving community-based chronic disease care: Cluster randomized trial evidence from Kenya. Soc Sci Med. 2024 Jun;351:116993. doi: 10.1016/j.socscimed.2024.116993. Epub 2024 May 17. PMID 38781744
- [Background] Liang A, Wilson-Barthes M, Galarraga O. Cost-effectiveness of differentiated care models that incorporate economic strengthening for HIV antiretroviral therapy adherence: a systematic review. Cost Eff Resour Alloc. 2024 May 24;22(1):46. doi: 10.1186/s12962-024-00557-w. PMID 38790050
- [Background] Vidal M. The Methodus medendi innovation in Giorgio Baglivi's work. Med Secoli. 2000;12(1):171-90. PMID 11624711
- [Background] Lyons C, Ching J, Tran DN, Kafu C, Wachira J, Koros H, Venkataramani M, Said J, Pastakia SD, Galarraga O, Genberg B. Social, economic and food insecurity among people living with HIV in Kenya during coinciding public health and environmental emergencies: a mixed-methods study. BMJ Public Health. 2024 Sep 23;2(2):e000836. doi: 10.1136/bmjph-2023-000836. eCollection 2024 Dec. PMID 40018611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1112 participants in 61 microfinance groups were screened for eligibility.
Pre-assignment Details: 900 participants in 57 microfinance groups were enrolled. An additional 300 participants not engaged in microfinance were frequency-matched and enrolled.
  We initially enrolled 1200 eligible participants in the study. We conducted randomization after (e.g., a few weeks following) enrollment to make community randomization more feasible. Between enrollment and randomization, n=45 participants left the study or were unable to be located, resulting in n=1155 participants ultimately randomized.
Units Other Than Participants: Microfinance Groups
Groups:
- Microfinance with Integrated, Community-based Care: Approximately half of enrolled microfinance groups will be randomized to receive the ICB intervention.
  Integrated Community-Based (ICB) Care: The intervention will be delivered quarterly during months 1-18 of the trial during regularly scheduled microfinance group meetings, and will include the following components: one-on-one consultation with a clinical officer in a private nearby location, distribution of antiretroviral therapy and other medications for diabetes and hypertension as needed, point-of-care laboratory testing if medically indicated, referrals to facilities for emergency or acute care needs, and group health education discussions.
  Microfinance: Group microfinance uses a client-driven model that involves community savings groups where members mobilize and manage their own savings, provide interest-bearing loans to group members, offer a limited form of financial insurance, and contribute to a social fund that is used for income-generating activities and in cases of emergency or welfare issues of group members.
  For this study, group microfinance will refer to existing, active AMPATH Group Integrated Savings for Empowerment (GISE) microfinance groups with a majority of group members who are AMPATH HIV patients and have disclosed their HIV status. Groups will be considered active if the group was formed at least 6 months prior to study baseline, is consistently meeting as scheduled, and is actively engaging in saving and loaning.
- Microfinance with Usual (Facility-based) Care: Approximately half of enrolled microfinance groups will be randomized to continue to receive usual chronic disease care from an AMPATH-supported rural health facility.
  Microfinance: Group microfinance uses a client-driven model that involves community savings groups where members mobilize and manage their own savings, provide interest-bearing loans to group members, offer a limited form of financial insurance, and contribute to a social fund that is used for income-generating activities and in cases of emergency or welfare issues of group members.
  For this study, group microfinance will refer to existing, active AMPATH Group Integrated Savings for Empowerment (GISE) microfinance groups with a majority of group members who are AMPATH HIV patients and have disclosed their HIV status. Groups will be considered active if the group was formed at least 6 months prior to study baseline, is consistently meeting as scheduled, and is actively engaging in saving and loaning.
- Usual (Facility-based) Care: A total of n=300 participants who receive usual care at an AMPATH health facility and who are not involved in microfinance will serve as frequency-matched, contemporaneous controls. These participants will be prospectively followed over the 18-months of the trial.
Period: Overall Study
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
Started | 407; 29 Microfinance Groups | 448; 28 Microfinance Groups | 300; 0 Microfinance Groups
Completed | 336; 29 Microfinance Groups | 381; 28 Microfinance Groups | 293; 0 Microfinance Groups
Not Completed | 71; 0 Microfinance Groups | 67; 0 Microfinance Groups | 7; 0 Microfinance Groups

BASELINE CHARACTERISTICS:
Population: The n=300 participants receiving usual (facility-based) care alone were not participating in a microfinance group, and were frequency-matched to the n=900 participants who were members of the n=57 enrolled microfinance groups.
Units Other Than Participants: Microfinance Groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care | Total
Number analyzed (Participants) | 407 | 448 | 300 | 1155
Number analyzed (Microfinance Groups) | 29 | 28 | 0 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.1) | 51.4 (11.7) | 52.6 (10.9) | 51.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 336 | 230 | 871
  Male | 102 | 112 | 70 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 407 | 448 | 300 | 1155
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 407 | 448 | 300 | 1155
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 407 | 448 | 300 | 1155

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 RNA Viral Load Suppression at 18-months
Description: Participants whose 18-month viral load assessment occurred before January 1, 2023 were considered suppressed if their viral load was <400 copies/mL. Following changes to Kenya's national HIV monitoring cutoffs that occurred during the trial, patients whose 18- month viral load assessment was on or after January 1, 2023 were considered suppressed if their viral load was <200 copies/mL.
Time Frame: 18 months
Population: Number of participants who provided a blood draw for viral load assessment (primary outcome) during their 18-month study visit. If a participant had a viral load result available in their medical record within the 3 months prior to their 18-month assessment date, then this result was used to assess their 18-month viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
Number analyzed (Participants) | 335 | 377 | 291
Participants | 326 | 365 | 275
Statistical Analysis 1: Comparison: Microfinance with Integrated, Community-based Care vs Microfinance with Usual (Facility-based) Care; For the primary outcome, the primary analysis was an intention-to-treat analysis that included all randomized participants comparing viral suppression at 18-months. Following studies of the effect of financial interventions, we powered the study to have at least 80% power to detect a 15% additive increase in viral suppression among microfinance group members receiving integrated community care compared to those receiving facility-based care, assuming 15% dropout; Test type: Superiority — Analysis of the primary outcome was conducted using a doubly-robust generalized estimating equation (GEE) with a logit link function. Multiple imputation was used to account for missing data on baseline covariates; Rubin's rule was used for variance estimation. The GEE model included the intervention arm, used an independence working correlation matrix and variance was estimated using a sandwich variance estimator for clustered data; p = 0.23, Wald test — Baseline values of variables (county, gender, age, education, income, viral load) were used for differential dropout adjustment for the primary comparison and differential dropout and confounding adjustments for comparisons to matched participants; Hypothesis: Microfinance with Integrated, Community-based Care > Microfinance with Usual Care in terms of viral suppression at 18-months; Odds Ratio, log = 0.84, 95% CI 2-sided [0.63 to 1.12] — The intervention effect was estimated using the log odds ratio coefficient associated with the intervention in the GEE. The primary hypothesis test of intervention effect was conducted using a Wald test and 95% Wald-based confidence intervals
Statistical Analysis 2: Comparison: Microfinance with Integrated, Community-based Care vs Usual (Facility-based) Care; A secondary analysis of the primary outcome included a comparison of viral suppression at 18- months, between each of the two randomized trial arms and the non-randomized, prospectively-followed, frequency-matched participants who were not engaged in microfinance. The secondary analysis used the same analytic model as the primary analysis, assuming no clustering in the non-randomized sample; Test type: Superiority; p < 0.001, Wald test — Hypothesis: Microfinance with Integrated, Community-based Care > Usual (Facility-based) Care in terms of viral suppression at 18-months; Odds Ratio, log = 2.16, 95% CI 2-sided [1.48 to 3.19]
Statistical Analysis 3: Comparison: Microfinance with Usual (Facility-based) Care vs Usual (Facility-based) Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.023, Wald test — Hypothesis: Microfinance with Usual (Facility-based) Care > Usual (Facility-based) Care in terms of viral suppression at 18-months; Odds Ratio, log = 1.42, 95% CI 2-sided [1.05 to 1.92]

2. Secondary Outcome: Retention in Care Each Quarter During 18-months of Follow-up
Description: A participant was considered retained in HIV care if they attended at least one HIV care visit in each quarter a visit was scheduled (always retained in care), where attending a visit was defined as attending a visit within +/- 28 days of their scheduled visit date (following AMPATH care protocols). Patients who had no visit(s) scheduled in a given quarter were considered retained for that quarter.
Time Frame: Between baseline and 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
Number analyzed (Participants) | 407 | 448 | 300
Participants | 315 | 235 | 51
Statistical Analysis 1: Comparison: Microfinance with Integrated, Community-based Care vs Microfinance with Usual (Facility-based) Care; The retention in care analysis was an intention-to-treat analysis that included all enrolled participants and used the same analysis methods as those for the viral suppression (primary outcome) analysis. The retention in care analyses were not adjusted for multiplicity and should be considered hypothesis generating; Test type: Superiority; p < 0.001, Wald test; Odds Ratio, log = 3.31, 95% CI 2-sided [2.58 to 4.26]
Statistical Analysis 2: Comparison: Microfinance with Integrated, Community-based Care vs Usual (Facility-based) Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Wald test; Odds Ratio, log = 7.51, 95% CI 2-sided [6.00 to 9.55]
Statistical Analysis 3: Comparison: Microfinance with Usual (Facility-based) Care vs Usual (Facility-based) Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Wald test; Odds Ratio, log = 2.56, 95% CI 2-sided [2.14 to 3.06]

3. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in systolic blood pressure (mm Hg) at 18 months as compared to baseline
Time Frame: Between baseline and 18 months
Population: This outcome was only measured for participants of randomized microfinance groups who provided a blood pressure reading at both baseline (month 0) and endline (month 18). Systolic blood pressure was not measured among frequency-matched usual care patients.
Measure: Mean (Standard Deviation); unit: mm Hg (millimeters of mercury)
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
Number analyzed (Participants) | 254 | 375 | 0
mm Hg (millimeters of mercury) | 0.25 (15.89) | 0.046 (14.26) |
Statistical Analysis 1: Comparison: Microfinance with Integrated, Community-based Care vs Microfinance with Usual (Facility-based) Care; Test type: Superiority; Wald test; Mean Difference (Final Values) = -0.206, 95% CI 2-sided [-2.595 to 2.183]

4. Secondary Outcome: Change in Random Blood Sugar (mmol/L)
Description: Change in random blood sugar (mmol/L) at 18 months as compared to baseline
Time Frame: Between baseline and 18 months
Population: Random blood sugar was only measured for participants of randomized microfinance groups who were clinically indicated to provide a blood glucose test at both baseline (month 0) and endline (month 18). Random blood sugar was not measured among frequency-matched usual care patients.
Measure: Mean (Standard Deviation); unit: mmol/L (millimoles per liter)
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
Number analyzed (Participants) | 232 | 346 | 0
mmol/L (millimoles per liter) | 0.276 (1.62) | -0.172 (1.45) |
Statistical Analysis 1: Comparison: Microfinance with Integrated, Community-based Care vs Microfinance with Usual (Facility-based) Care; Test type: Superiority; Wald test; Mean Difference (Final Values) = -0.4478, 95% CI 2-sided [-0.701 to -0.194]

ADVERSE EVENTS:
Time Frame: 18 months
Description: During the 18-month trial, our investigative team followed all procedures outlined in the Protection of Human Subjects Section of the Overall Project Protocol. No adverse events related to the study intervention occurred during the trial. All deaths that occurred during the trial were unrelated to the intervention or to study procedures, and were reported to the IRB of record (Moi University) within the required time frame.
Groups:
- Microfinance with Integrated, Community-based Care: Half of enrolled microfinance groups with approximately n=450 participants will be randomized to receive the ICB intervention.
  Integrated Community-Based (ICB) Care: The intervention will be delivered quarterly during months 1-18 of the trial during regularly scheduled microfinance group meetings, and will include the following components: one-on-one consultation with a clinical officer in a private nearby location, distribution of antiretroviral therapy and other medications for diabetes and hypertension as needed, point-of-care laboratory testing if medically indicated, referrals to facilities for emergency or acute care needs, and group health education discussions.
  Microfinance: Group microfinance uses a client-driven model that involves community savings groups where members mobilize and manage their own savings, provide interest-bearing loans to group members, offer a limited form of financial insurance, and contribute to a social fund that is used for income-generating activities and in cases of emergency or welfare issues of group members.
  For this study, group microfinance will refer to existing, active AMPATH Group Integrated Savings for Empowerment (GISE) microfinance groups with a majority of group members who are AMPATH HIV patients and have disclosed their HIV status. Groups will be considered active if the group was formed at least 6 months prior to study baseline, is consistently meeting as scheduled, and is actively engaging in saving and loaning.
- Microfinance with Usual (Facility-based) Care: Half of enrolled microfinance groups with approximately n=450 participants will be randomized to continue to receive usual chronic disease care from an AMPATH-supported rural health facility.
  Microfinance: Group microfinance uses a client-driven model that involves community savings groups where members mobilize and manage their own savings, provide interest-bearing loans to group members, offer a limited form of financial insurance, and contribute to a social fund that is used for income-generating activities and in cases of emergency or welfare issues of group members.
  For this study, group microfinance will refer to existing, active AMPATH Group Integrated Savings for Empowerment (GISE) microfinance groups with a majority of group members who are AMPATH HIV patients and have disclosed their HIV status. Groups will be considered active if the group was formed at least 6 months prior to study baseline, is consistently meeting as scheduled, and is actively engaging in saving and loaning.
- Usual (Facility-based) Care: n=300 participants who receive usual care at an AMPATH health facility and who are not involved in microfinance will serve as frequency-matched, contemporaneous controls. These participants will be prospectively followed over the 18-months of the trial.
Arm/Group | Microfinance with Integrated, Community-based Care | Microfinance with Usual (Facility-based) Care | Usual (Facility-based) Care
All-Cause Mortality (participants affected / at risk) | 3/407 | 2/448 | 0/300
Serious Adverse Events (participants affected / at risk) | 3/407 | 2/448 | 0/300
Other Adverse Events (participants affected / at risk) | 0/407 | 0/448 | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microfinance with Integrated, Community-based Care (N=407) | Microfinance with Usual (Facility-based) Care (N=448) | Usual (Facility-based) Care (N=300)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Participant was an enrolled microfinance group member receiving usual (facility-based) care. Participant died during study follow up due to cervical cancer. Their death was determined not to be associated with the research.
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) — Participant was an enrolled microfinance group member receiving usual (facility-based) care. Participant died during study follow up due to unknown causes. Their death was determined not to be associated with the research.
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Participant was an enrolled microfinance group member receiving integrated community-based care. Participant died during study follow up due to suspected esophageal malignancy. Their death was determined not to be associated with the research.
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Participant was an enrolled microfinance group member receiving integrated community-based care. Participant died during study follow up due to stroke. Their death was determined not to be associated with the research.
Death (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Participant was an enrolled microfinance group member receiving integrated community-based care. Participant died during study follow up due to pneumonia. Their death was determined not to be associated with the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Updated Project Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT04417127/Prot_SAP_ICF_000.pdf